CLINICAL TRIAL: NCT06157034
Title: Prokinetic Effect of Selected Nutraceuticals on Management of Gastrointestinal Disturbances Among Pulmonary Tuberculosis Patients
Brief Title: Prokinetic Effect of Selected Nutraceuticals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Open University Islamabad (Other)
Responsible Party: Principal Investigator, Asma Latif, Dietician, Allama Iqbal Open University Islamabad
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Allama Iqbal Open University.
Record Dates: First submitted 2020-11-01; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pulmonary Tuberculosis; Gastro-Intestinal Disorder
MeSH Terms: conditions — Tuberculosis, Pulmonary; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Phase1 - 200 population size will be divided into 4 treatment groups
  Phase2
  * The phase will check the impact of selected nutraceuticals on TB patients with dietary counseling and all collected data in Phase1 will be repeated at the end
  * 3 selected nutraceuticals Zingiber officinale, Carum carvi, and Mentha spicata will be used against placebo and each placed in a separate group with 50 subjects for 3 months
  * Before dispensing treatments, raw material will be processed and encapsulated in prescribed doses in 4 groups after breakfast and dinner T1-Placebo 100mg/d, T2-Zingiber Officinale powder (500mg 2x/d=1000mg/d), T3-Carum powder(1g 2x/d=2g/d), T4-Mentha oil(2% of oil1.5ml 2x/d=30mg/d)
  Phase3
  - The impact of withholding the intervention will be studied to observe any change in selected parameters
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Exploratory (No Intervention): * After sampling the study population of 200 will be divided into four (04) treatment groups i.e. T1 (Placebo), T2 (Zingiber officinale), T3 (Carum carvi, L), and T4 (Mentha spicata L).
  * Each group will be allotted 50 subjects
- T1 (Experimental): * In the pursuit of scientific understanding, clinical studies play a pivotal role in evaluating the efficacy of treatments. One essential aspect is the inclusion of a placebo group, denoted as the T1 group in this study. Participants in this group will be administered inert material in the form of 100 mg capsules, serving as a baseline for comparison against the active treatment groups.
  * Group Designation: T1 Placebo Group
    * Intervention: 100 mg capsule containing inert material
    * Dosage Frequency: Daily
    * Duration: 3 months
    * Number of Participants: 50 subjects
  * Participants in the T1 Placebo Group are fully informed about the nature of the study, including the possibility of receiving a placebo.
  * Informed consent is obtained from each participant, ensuring that they are aware of the study's objectives and the potential for receiving an inactive treatment.
  Interventions: Other: Placebo
- T2 (Experimental): * Zingiber officinale, commonly known as ginger, has been of interest for its potential health benefits.
  * In this clinical study, the T2 treatment group is designated to receive Zingiber officinale powder.
  * Intervention Details:
    * Group Designation: T2 Treatment Group
    * Intervention: Zingiber officinale powder
    * Dosage: 500 mg capsules
    * Dosage Frequency: Twice daily
    * Total Daily Dosage: 1000 mg
    * Administration Timing: After breakfast and dinner
    * Duration: 3 months
  * Throughout the study duration, data will be systematically collected from participants in the T3 treatment group. This data may include subjective reports, clinical assessments, and laboratory analyses.
  Interventions: Dietary Supplement: Zingier officinale powder
- T3 (Experimental): * Carum carvi, L, commonly known as caraway, is a botanical with a rich history of traditional use. In this clinical study, a treatment group, denoted as T3, is established to investigate the effects of encapsulated Carum carvi, L powder in alleviating the gastrointestinal disturbances among TB patients.
  * Intervention Details:
    * Generic Name: Carum carvi, L powder
    * Dosage Form: Encapsulated
    * Dosage: 1 g per capsule
    * Frequency: Twice daily
    * Total Daily Dosage: 2 g/day
    * Administration Timing: After breakfast and dinner
    * Duration of Treatment: 3 months
  * Throughout the study duration, data will be systematically collected from participants in the T3 treatment group. This data may include subjective reports, clinical assessments, and laboratory analyses.
  Interventions: Dietary Supplement: Carum carvi, L powder
- T4 (Experimental): * Mentha spicata L, commonly known as spearmint, is renowned for its aromatic properties and potential health benefits. In this clinical study, a treatment group, designated as T4, is established to explore the effects of encapsulated Mentha spicata oil.
  * Intervention Details:
    * Generic Name: Mentha spicata oil
    * Dosage Form: Encapsulated
    * Concentration: 2% of Spearmint essential oil
    * Dosage: 1.5 ml per capsule
    * Frequency: Twice daily
    * Total Daily Dosage: 30 ml/day
    * Administration Timing: After breakfast and dinner
    * Duration of Treatment: 3 months
  * Throughout the study duration, data will be systematically collected from participants in the T4 treatment group. This data may include subjective reports, clinical assessments, and laboratory analyses.
  Interventions: Dietary Supplement: Mentha spicata oil
- Washout period (No Intervention): * In this phase impact of withholding the intervention on all parameters will be studied.
  * All parameters included in phase1 and 2 will be repeated after one month accordingly, to observe any change in selected parameters after discontinuation of intervention.

INTERVENTIONS:
Other: Placebo — Inert Material
  Arms: T1
Dietary Supplement: Zingier officinale powder — The raw form of Zingiber officinale will be grounded in powder by manual grinding and will be encapsulated.
  Arms: T2
Dietary Supplement: Carum carvi, L powder — The raw form of Carum carvi, L will be grounded in powder by manual grinding and will be encapsulated.
  Arms: T3
Dietary Supplement: Mentha spicata oil — Mentha spicata L will be extracted in the form of oil and will be encapsulated.
  Arms: T4

SUMMARY:
Anti-Tuberculosis Treatment (ATT) is one of the effective treatments of tuberculosis but the use of drugs for a long time put an adverse effect on the gut and other organs of the body. Nutraceuticals are the cheapest natural sources with therapeutic effects. These natural medicines help in alleviating gastrointestinal disturbances. This study will be conducted to overcome gastrointestinal issues with the help of nutraceuticals, which are more acceptable by the majority and have no side effects.

DETAILED DESCRIPTION:
The aim of this study will be to evaluate if Zingiber officinale, Carum carvi, L, and Mentha spicata L nutraceuticals can help in alleviating gastrointestinal disturbances in subjects which are more acceptable by the majority and have no side effects.

This Randomized Control interventional three arms Trial will comprise three phases. Patients will be randomized to Zingiber officinale, Carum carvi, L, and Mentha spicata L nutraceuticals or placebo for three months. We will evaluate symptoms assessment, dietary assessment, biochemical and physical analysis i.e. Acid-Fast Bacillus (AFB) for sputum, Chest X-ray (CXR), and Complete Blood Count (CBC) at baseline and after 3 months since the study started.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Pulmonary TB patients (both genders)
* Age group 18-65 years
* Symptoms criteria (Rome IV)

Exclusion Criteria:

* Patients ˃ 18 years and ˂ 65 years.
* Patients registered with extra pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
--GIT disturbances | "1 Month" at study commencement (Phase 1)
  GIT disturbences will be assessed through ROME IV including abdominal pain, bloating, vomiting and nausea in Phase 1.
GIT disturbances | Termination of Phase 2 (Intervention period) "3 Months"
  GIT disturbences will be assessed through ROME IV including abdominal pain, bloating, vomiting and nausea in Phase 2 after completion of three-month intervention.
GIT disturbances | Termination of phase 3 (Washout period) "1 Month"
  GIT disturbences will be assessed through ROME IV including abdominal pain, bloating, vomiting and nausea in Phase 3 which is wash out time.

SECONDARY OUTCOMES:
Body Mass Index | "through study completion, an average of 9 months"
  Measurements will be taken in triplicate. Height will be measured to the nearest 0.5 cm with a stadiometer (or knee height, ulnar length or arm span [demispan] for those persons unable to stand fully erect); body weight will be measured to the nearest 0.1 kg.
A self-designed / pretested questionnaire | "through study completion, an average of 9 months"
  will be used to collect data on other determinants that affect patients regarding disease history, and dietary history. Agarwal Socio-economic status (SES) performa will be used.
Acid-Fast Bacillus (sputum) | "through study completion, an average of 9 months"
  sample will be taken at time of enrollment in study to make diagnosis of Tuberculosis
Chest X-ray (CXR) | "1 Day" at study commencement (Phase 1)
  Phase 1 in which subjects will be enrolled and their CXR will be taken as criteria for diagnosis of TB
Complete blood count (CBC) | "1 Day" at study commencement (Phase 1)
  Phase 1 in which subjects will be enrolled and their CBC will be taken as criteria for diagnosis of TB

CONTACTS AND LOCATIONS:
Overall Officials: Asma Latif, PhD Scholar, Principal Investigator — Sheikh Zaid Medical / college.Rahim Yar Khan.Pakistan
Locations (1):
- Sheikh Zayed Medical / college, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No